CLINICAL TRIAL: NCT06959368
Title: A Randomised Controlled Trial Comparing Vonoprazan Triple Therapy (Vonoprazan, Amoxicillin, Clarithromycin), and Standard Triple Therapy (Esomeprazole, Amoxicillin, Clarithromycin) for Helicobacter Pylori Eradication in Indian Population. VECTOR Trial - Vonoprazan Evaluation Compared to Standard Triple Therapy in Helicobacter Pylori eRadication
Brief Title: Vonoprazan Evaluation Compared to Standard Triple Therapy in Helicobacter Pylori eRadication
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VECTOR-01
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-02

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Esomeprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vonoprazan triple therapy (Active Comparator): • Vonoprazan Triple Therapy: Vonoprazan 20 mg, Amoxicillin 1 g, Clarithromycin 500 mg (all twice daily).
  Interventions: Drug: Vonoprazan 20mg, Esomeprazole 40 mg, Amoxicillin 1 g, Clarithromycin 500 mg
- Standard triple therapy (Active Comparator): • Standard Triple Therapy: Esomeprazole 40 mg, Amoxicillin 1 g, Clarithromycin 500 mg (all twice daily).
  Interventions: Drug: Vonoprazan 20mg, Esomeprazole 40 mg, Amoxicillin 1 g, Clarithromycin 500 mg

INTERVENTIONS:
Drug: Vonoprazan 20mg, Esomeprazole 40 mg, Amoxicillin 1 g, Clarithromycin 500 mg — Participants will receive the respective drug regimens twice daily. The Vonoprazan triple therapy arm will administer Vonoprazan 20 mg, Amoxicillin 1 g, and Clarithromycin 500 mg twice daily. The Standard triple therapy arm will administer Esomeprazole 40 mg, Amoxicillin 1 g, and Clarithromycin 500 mg twice daily.

SUMMARY:
Helicobacter pylori (H Pylori) infection is associated with functional dyspepsia, peptic ulcer disease, atrophy and gastric cancer. The bacterium has been classified as grade I carcinogen by the WHO in 1994(1). Based on the clinical and microbiological data it is now well known to be the strongest risk factor for developing intestinal type and diffuse type of adenocarcinoma(2-4). While testing and treating asymptomatic persons is a grey area, it is now recommended to rule out H. pylori in un-investigated dyspepsia patients (5-7), and if detected, it must be treated. However, worldwide and especially in the Asian countries, we face a widespread problem of antibiotic resistance(8,9). Regimens are typically selected based on the varying regional clarithromycin resistance(6,9). There is a need for an efficient and reliable empirical therapy that can be universal, has maximal eradication rates irrespective of resistance patterns, has good compliance and minimal adverse events without the emergence of superbugs. We also need a reliable rescue therapy for H. pylori eradication failure.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years - 80 years)
* Patient visiting clinic with dyspepsia, GERD, or non-bleeding peptic ulcer
* 13C-urea breath test (UBT) positive/ Rapid urease test positive (RUT) on endoscopic biopsy
* Off PPIs for 2 weeks

Exclusion Criteria:

* Penicillin allergy
* Recent use of antibiotics in the past 1 month
* Previous H. pylori therapy
* Intestinal metaplasia, gastric cancer, bleeding peptic ulcer
* Patient who is unable to understand study protocol or not consenting
* Pregnancy, lactation
* Patient on anticoagulation, NSAIDs
* Patient using drugs with interactions with vonoprazan, amoxicillin, clarithromycin or PPIs
* Cirrhosis, Chronic kidney disease, chronic lung disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
A randomised controlled trial comparing Vonoprazan triple therapy (Vonoprazan, Amoxicillin, Clarithromycin), and standard triple therapy (Esomeprazole, Amoxicillin, Clarithromycin) for Helicobacter pylori eradication in Indian population. VECTOR trial | 1 year
  The primary outcome measurement is to assess the eradication of H. pylori i.e. negative UBT or stool antigen test 4 weeks after treatment

SECONDARY OUTCOMES:
Assessment of adverse events and eradication rates in antibiotic-resistant strains. | 1 year
  Assessment of adverse events and eradication rates in antibiotic-resistant strains.

CONTACTS AND LOCATIONS:
Locations (1):
- AIG hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No